CLINICAL TRIAL: NCT02790749
Title: Periacetabular Osteotomy With Versus Without Adjunctive Hip Arthroscopy for Intra-Articular Pathology in Hip Dysplasia: a Prospective Randomized Trial
Brief Title: Periacetabular Osteotomy With Versus Without Adjunctive Hip Arthroscopy
Acronym: PRSPAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Michael Muldoon, M.D., Staff Physician, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1603903
Record Dates: First submitted 2016-05-18; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Hip Dysplasia
Keywords: Developmental hip dysplasia; Intra-articular pathology; Adult hip dysplasia; Labral tear, hip; Chondromalacia, hip
MeSH Terms: conditions — Hip Dislocation; Developmental Dysplasia of the Hip; Cartilage Diseases | interventions — Polyamine Oxidase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAO with adjunctive hip arthroscopy (Experimental): Patients undergoing periacetabular osteotomy (PAO) with adjunctive hip arthroscopy.
  Interventions: Procedure: Adjunctive hip arthroscopy to accompany PAO
- PAO WITHOUT adjunctive hip arthroscopy (Active Comparator): Patients undergoing periacetabular osteotomy (PAO) WITHOUT adjunctive hip arthroscopy.
  Interventions: Procedure: PAO without adjunctive hip arthroscopy

INTERVENTIONS:
Procedure: Adjunctive hip arthroscopy to accompany PAO — This is the experimental group: those patients who undergo adjunctive hip arthroscopy in addition to periacetabular osteotomy (PAO).
  Arms: PAO with adjunctive hip arthroscopy
Procedure: PAO without adjunctive hip arthroscopy — This is the control group: those patients who undergo periacetabular osteotomy (PAO) alone, without adjunctive hip arthroscopy.
  Arms: PAO WITHOUT adjunctive hip arthroscopy

SUMMARY:
Although evidence is amassing regarding the role of intra-articular pathology in the surgical management of adolescents and adults with hip dysplasia, the optimal method of detection and especially management of this pathology remains unclear. No studies exist to compare clinical outcomes and hip survival between arthroscopy and arthrotomy in patients with mechanical hip pain undergoing periacetabular osteotomy (PAO) for dysplasia, and this is what the investigators aim to achieve in the current prospective randomized surgical trial.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip is an increasingly well-recognized problem in adolescents, young adults, and middle-age adults. Surgical correction with periacetabular osteotomy (PAO) gives good results at moderate-term follow-up, according to recent studies. Increasingly recognized also is the presence of intra-articular sources of hip pain in these patients, such as cartilage disease and labral pathology. These can manifest as certain clinical and radiologic findings pre-operatively. However, the role of operative management of these problems, and specifically the role of arthroscopy, remains unclear. Historically, intra-articular pathology in patients with dysplasia has been managed with open incision of the joint capsule (arthrotomy) toward the end of the PAO procedure. However, recent evidence suggests that this open arthrotomy may be missing the detection of subtle intra-articular pathology and that arthroscopy immediately prior to PAO, under the same anesthetic, may be a safe and highly effective management strategy. The exact clinical implications of these subtle findings are not yet clear.

In this prospective randomized comparative effectiveness study, the investigators aim to compare clinical and surgical outcomes measures including rates of reoperation and the patient reported outcomes measures (PROMs) non-arthritic hip score (NAHS), Hip Outcome Score (HOS), modified Harris Hip Score (mHHS), iHOT-12 score, between two groups of patients (N=22 per parallel arm) undergoing PAO for dysplasia: those randomized to arthroscopy with PAO versus those randomized to PAO alone.

The investigators aim to elucidate the degree of clinical benefit of improved detection and management of intra-articular pathology afforded by arthroscopy versus PAO with arthrotomy alone at follow-up of a minimum of one year. Rates of reoperation and PROMs will be assessed at one year post-operatively and at the conclusion of the study two years after enrollment of the first patient. PROMs will also be assessed at 3 and 6 months post-operatively to allow repeated-measures analysis in measuring improvement from pre-operative values.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 50
* Moderate or severe dysplasia by radiographic parameters
* Physical examination and/or MR arthrography consistent with intra-articular pathology (equivocal or even negative MR arthrogram for labral tear, chondral flap, ligamentum teres tear, or osteochondral defect, is not grounds for exclusion, since broadly spaced "cuts" of MR imaging may miss small tears)
* English- or Spanish-speaking
* signed written informed consent for surgery and for research prior to surgery

Exclusion Criteria:

* Tönnis grade II or III arthritis at baseline
* MR cartilage imaging indicating severe arthritis
* Prior surgery on the same hip
* Contralateral lower limb pathology that threatens validity of outcomes measures directed at the operative hip
* History of thromboembolic disease in the lower extremity, pulmonary embolus, or pre-existing thrombophilic blood disorder
* Inability to participate in or comply with appropriate rehabilitation protocols
* Inability to comprehend and follow instructions, or mental incapacity barring consent
* Pregnant women
* Lost to follow-up before one year, unless total hip replacement performed before one year (then included for survival analysis)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of reoperation by final follow-up | One year
  Incidence of repeat arthroscopy due to persistent mechanical symptoms after index PAO
NAHS (non-arthritic hip score) | One year
  Absolute value of, and measure of post-operative improvement in, validated questionnaire known as NAHS--Non-Arthritic Hip Score

SECONDARY OUTCOMES:
iHOT-12: 12-question version of the international Hip Outcome Tool | one year
  questionnaire known as iHOT-12: the 12-question version of the international Hip Outcome Tool
HOS: Hip Outcome Score | one year
  questionnaire known as the HOS: Hip Outcome Score
mHHS: Modified Harris Hip Score | one year
  questionnaire known as mHHS: Modified Harris Hip Score

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Muldoon, MD, Principal Investigator — Sharp HealthCare

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ganz R, Leunig M, Leunig-Ganz K, Harris WH. The etiology of osteoarthritis of the hip: an integrated mechanical concept. Clin Orthop Relat Res. 2008 Feb;466(2):264-72. doi: 10.1007/s11999-007-0060-z. Epub 2008 Jan 10. PMID 18196405
- [Background] Klaue K, Durnin CW, Ganz R. The acetabular rim syndrome. A clinical presentation of dysplasia of the hip. J Bone Joint Surg Br. 1991 May;73(3):423-9. doi: 10.1302/0301-620X.73B3.1670443.
- [Background] Siebenrock KA, Scholl E, Lottenbach M, Ganz R. Bernese periacetabular osteotomy. Clin Orthop Relat Res. 1999 Jun;(363):9-20. PMID 10379300
- [Background] Ganz R, Klaue K, Vinh TS, Mast JW. A new periacetabular osteotomy for the treatment of hip dysplasias. Technique and preliminary results. Clin Orthop Relat Res. 1988 Jul;(232):26-36. PMID 3383491
- [Background] Steppacher SD, Tannast M, Ganz R, Siebenrock KA. Mean 20-year followup of Bernese periacetabular osteotomy. Clin Orthop Relat Res. 2008 Jul;466(7):1633-44. doi: 10.1007/s11999-008-0242-3. Epub 2008 May 1. PMID 18449617
- [Background] Kemp JL, Collins NJ, Makdissi M, Schache AG, Machotka Z, Crossley K. Hip arthroscopy for intra-articular pathology: a systematic review of outcomes with and without femoral osteoplasty. Br J Sports Med. 2012 Jul;46(9):632-43. doi: 10.1136/bjsports-2011-090428. Epub 2011 Dec 22. PMID 22194221
- [Background] Clohisy JC, Schutz AL, St John L, Schoenecker PL, Wright RW. Periacetabular osteotomy: a systematic literature review. Clin Orthop Relat Res. 2009 Aug;467(8):2041-52. doi: 10.1007/s11999-009-0842-6. Epub 2009 Apr 21. PMID 19381741
- [Background] Davey JP, Santore RF. Complications of periacetabular osteotomy. Clin Orthop Relat Res. 1999 Jun;(363):33-7. PMID 10379302
- [Background] Thawrani D, Sucato DJ, Podeszwa DA, DeLaRocha A. Complications associated with the Bernese periacetabular osteotomy for hip dysplasia in adolescents. J Bone Joint Surg Am. 2010 Jul 21;92(8):1707-14. doi: 10.2106/JBJS.I.00829. PMID 20660233
- [Background] Ginnetti JG, Pelt CE, Erickson JA, Van Dine C, Peters CL. Prevalence and treatment of intraarticular pathology recognized at the time of periacetabular osteotomy for the dysplastic hip. Clin Orthop Relat Res. 2013 Feb;471(2):498-503. doi: 10.1007/s11999-012-2602-2. PMID 23054510
- [Background] Muldoon MP, Santore RF. Abstract presented at Western Orthopedic Association. Adjunctive Hip Arthroscopy with Periacetabular Osteotomy for Hip Dysplasia. 2007.
- [Background] Fujii M, Nakashima Y, Noguchi Y, Yamamoto T, Mawatari T, Motomura G, Iwamoto Y. Effect of intra-articular lesions on the outcome of periacetabular osteotomy in patients with symptomatic hip dysplasia. J Bone Joint Surg Br. 2011 Nov;93(11):1449-56. doi: 10.1302/0301-620X.93B11.27314. PMID 22058293
- [Background] Domb BG, LaReau J, Redmond JM. Combined hip arthroscopy and periacetabular osteotomy: indications, advantages, technique, and complications. Arthrosc Tech. 2014 Jan 10;3(1):e95-e100. doi: 10.1016/j.eats.2013.09.002. eCollection 2014 Feb. PMID 24843847
- [Background] Ginnetti JG, Erickson J, Peters CL. Periacetabular osteotomy: intra-articular work. Instr Course Lect. 2013;62:279-86. PMID 23395033
- [Background] Ross JR, Zaltz I, Nepple JJ, Schoenecker PL, Clohisy JC. Arthroscopic disease classification and interventions as an adjunct in the treatment of acetabular dysplasia. Am J Sports Med. 2011 Jul;39 Suppl:72S-8S. doi: 10.1177/0363546511412320. PMID 21709035
- [Background] Nassif NA, Schoenecker PL, Thorsness R, Clohisy JC. Periacetabular osteotomy and combined femoral head-neck junction osteochondroplasty: a minimum two-year follow-up cohort study. J Bone Joint Surg Am. 2012 Nov 7;94(21):1959-66. doi: 10.2106/JBJS.K.01038. PMID 23138238
- [Background] Peters CL, Sierra RJ; Session Participants. Report of breakout session: Intraarticular work during periacetabular osteotomy--simultaneous arthrotomy or hip arthroscopy? Clin Orthop Relat Res. 2012 Dec;470(12):3456-8. doi: 10.1007/s11999-012-2414-4. No abstract available. PMID 22723243
- [Background] McCarthy JC. The diagnosis and treatment of labral and chondral injuries. Instr Course Lect. 2004;53:573-7. PMID 15116646
- [Background] Martin RL, Irrgang JJ, Sekiya JK. The diagnostic accuracy of a clinical examination in determining intra-articular hip pain for potential hip arthroscopy candidates. Arthroscopy. 2008 Sep;24(9):1013-8. doi: 10.1016/j.arthro.2008.04.075. Epub 2008 Jun 16. PMID 18760208
- [Background] Redmond JM, Gupta A, Stake CE, Domb BG. The prevalence of hip labral and chondral lesions identified by method of detection during periacetabular osteotomy: arthroscopy versus arthrotomy. Arthroscopy. 2014 Mar;30(3):382-8. doi: 10.1016/j.arthro.2013.11.013. Epub 2014 Jan 22. PMID 24461141
- [Background] Peters CL, Erickson JA, Anderson MB, Anderson LA. Preservation of the rectus femoris origin during periacetabular osteotomy does not compromise acetabular reorientation. Clin Orthop Relat Res. 2015 Feb;473(2):608-14. doi: 10.1007/s11999-014-3837-x. PMID 25091227
- [Background] Papavasiliou AV, Bardakos NV. Complications of arthroscopic surgery of the hip. Bone Joint Res. 2012 Jul 1;1(7):131-44. doi: 10.1302/2046-3758.17.2000108. Print 2012 Jul. PMID 23610683
- [Background] Sambandam SN, Hull J, Jiranek WA. Factors predicting the failure of Bernese periacetabular osteotomy: a meta-regression analysis. Int Orthop. 2009 Dec;33(6):1483-8. doi: 10.1007/s00264-008-0643-7. Epub 2008 Aug 22. PMID 18719916
- [Background] Matheney T, Kim YJ, Zurakowski D, Matero C, Millis M. Intermediate to long-term results following the bernese periacetabular osteotomy and predictors of clinical outcome: surgical technique. J Bone Joint Surg Am. 2010 Sep;92 Suppl 1 Pt 2:115-29. doi: 10.2106/JBJS.J.00646. PMID 20844169
- [Background] Soderman P, Malchau H. Is the Harris hip score system useful to study the outcome of total hip replacement? Clin Orthop Relat Res. 2001 Mar;(384):189-97. doi: 10.1097/00003086-200103000-00022. PMID 11249165
- [Background] Clohisy JC, Carlisle JC, Beaule PE, Kim YJ, Trousdale RT, Sierra RJ, Leunig M, Schoenecker PL, Millis MB. A systematic approach to the plain radiographic evaluation of the young adult hip. J Bone Joint Surg Am. 2008 Nov;90 Suppl 4(Suppl 4):47-66. doi: 10.2106/JBJS.H.00756. No abstract available. PMID 18984718
- [Background] Bond JL, Knutson ZA, Ebert A, Guanche CA. The 23-point arthroscopic examination of the hip: basic setup, portal placement, and surgical technique. Arthroscopy. 2009 Apr;25(4):416-29. doi: 10.1016/j.arthro.2008.08.021. Epub 2008 Nov 22. PMID 19341931
- [Background] Nunley RM, Prather H, Hunt D, Schoenecker PL, Clohisy JC. Clinical presentation of symptomatic acetabular dysplasia in skeletally mature patients. J Bone Joint Surg Am. 2011 May;93 Suppl 2:17-21. doi: 10.2106/JBJS.J.01735. PMID 21543683
- [Background] Burnett RS, Della Rocca GJ, Prather H, Curry M, Maloney WJ, Clohisy JC. Clinical presentation of patients with tears of the acetabular labrum. J Bone Joint Surg Am. 2006 Jul;88(7):1448-57. doi: 10.2106/JBJS.D.02806. PMID 16818969
- [Background] Thorborg K, Tijssen M, Habets B, Bartels EM, Roos EM, Kemp J, Crossley KM, Holmich P. Patient-Reported Outcome (PRO) questionnaires for young to middle-aged adults with hip and groin disability: a systematic review of the clinimetric evidence. Br J Sports Med. 2015 Jun;49(12):812. doi: 10.1136/bjsports-2014-094224. Epub 2015 Jan 13. PMID 25586913
- [Background] Griffin DR, Parsons N, Mohtadi NG, Safran MR; Multicenter Arthroscopy of the Hip Outcomes Research Network. A short version of the International Hip Outcome Tool (iHOT-12) for use in routine clinical practice. Arthroscopy. 2012 May;28(5):611-6; quiz 616-8. doi: 10.1016/j.arthro.2012.02.027. PMID 22542434
- [Background] Harris JD, McCormick FM, Abrams GD, Gupta AK, Ellis TJ, Bach BR Jr, Bush-Joseph CA, Nho SJ. Complications and reoperations during and after hip arthroscopy: a systematic review of 92 studies and more than 6,000 patients. Arthroscopy. 2013 Mar;29(3):589-95. doi: 10.1016/j.arthro.2012.11.003. PMID 23544691
- [Background] Bedi A, Chen N, Robertson W, Kelly BT. The management of labral tears and femoroacetabular impingement of the hip in the young, active patient. Arthroscopy. 2008 Oct;24(10):1135-45. doi: 10.1016/j.arthro.2008.06.001. PMID 19028166